CLINICAL TRIAL: NCT06392906
Title: Orbital Radiotherapy in Grave's Ophthalmopathy 1 Week vs 2 Weeks: A Phase II Randomized Controlled Trial (OraGO-1 Trial)
Brief Title: Orbital Radiotherapy in Grave's Ophthalmopathy 1 Week vs 2 Weeks (OraGO-1 Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janjira Petsuksiri (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor-Investigator, Janjira Petsuksiri, Associate Professor Doctor, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI208/2024
Record Dates: First submitted 2024-03-30; First posted 2024-05-01 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Associated Ophthalmopathy
Keywords: radiation therapy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Intervention Model Description: Phase 2 randomized control trial comparing between standard radiation therapy arm (20 Gy in 10 fractions) and experimental radiation therapy arm (10 Gy in 5 fractions)
Masking Description: In this study, both participants and researchers are aware of the treatment administered due to the necessity for close monitoring of treatment outcomes and side effects by radiation oncologists and ophthalmologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 week external beam radiation therapy (Experimental): 10 Gy in 5 fractions of external beam radiation therapy
  Interventions: Radiation: Short course radiation therapy
- 2 week external beam radiation therapy (Active Comparator): 20 Gy in 10 fractions of standard fraction external beam radiation therapy
  Interventions: Radiation: Standard course radiation therapy

INTERVENTIONS:
Radiation: Short course radiation therapy — 5 daily radiation treatments
  Other Names: 10 Gy in 5 fractions of radiation therapy
  Arms: 1 week external beam radiation therapy
Radiation: Standard course radiation therapy — 10 daily radiation treatments
  Other Names: 20 Gy in 10 fractions of radiation therapy
  Arms: 2 week external beam radiation therapy

SUMMARY:
Thyroid ophthalmopathy, also known as thyroid eye disease or Graves' ophthalmopathy, is a condition characterized by inflammation and swelling of the tissues around the eyes, often accompanied by protrusion of the eyeballs. This condition can lead to significant discomfort, visual disturbances, and in severe cases, permanent vision loss.

Primary treatment modalities are intravenous methylprednisolone (IVMP) and other medications for patients with moderate to severe and active thyroid eye disease. In addition, external beam radiation therapy (ERT) is an another treatment option in combination with IVMP.

Radiation therapy delivers targeted doses of ionizing radiation to the affected orbital tissues, effectively reducing inflammation. This approach is particularly beneficial for patients who may not respond adequately to steroid therapy alone or those who experience recurrent disease flares.

This study will test the efficacy of a shortened treatment regimen comprising 5 sessions of ERT to a standard protocol of 10 treatments. The primary aim is to ascertain the effectiveness of shorted radiation treatment while improving patients' quality of life.

DETAILED DESCRIPTION:
The research methodology of this study involves comparing the standard protocol of 10 radiation treatments with a modified approach comprising 5 treatments of daily External Beam Radiation Therapy (ERT).

The primary objective of this investigation is to assess whether reducing the number of radiation treatments while maintaining the effectiveness of the therapy can lead to improvements in the quality of life for patients with thyroid ophthalmopathy.

By comparing these two treatment regimens, researchers aim to evaluate the efficacy and safety of the abbreviated radiation schedule in managing the symptoms and progression of the disease.

Participants enrolled in the study will be randomized into two groups: one receiving the standard 10 treatments and the other receiving the modified 5-treatment regimen of daily ERT. Throughout the study period, participants will undergo comprehensive assessments to monitor changes in symptoms, vision, and quality of life. These evaluations will include ophthalmic examinations, imaging studies, and patient-reported outcome measures to capture both objective and subjective measures of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patient with active moderate to severe thyroid eye disease with a CAS > 4 with/ without diplopia before starting IVMP
* Patient with poor response to 3 doses of IVMP (CAS drop < 1) หรือ CAS score > 3 after 3 doses of IVMP
* Patients with diplopia after 3 doses of IVMP
* Patients with Graves' Ophthalmopathy who have maintained euthyroidism
* Non-pregnant adults (aged 35 years or older)

Exclusion Criteria:

* Individuals with severe hypertension or diabetic retinopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Activity Score (CAS) change | 6 months after initiation of IVMP
  To evaluate the non-inferiority of outcomes in terms of the patient's proportion of converting from active (CAS > 4) to inactive eye disease (CAS <3) with CAS drop > 2 points, following orbital radiotherapy in combination with IVMP, comparing standard and reduced-dose orbital radiotherapy
  CAS score range from 1-7, initially and range from 1-10 at 1-3 months follow-up period. Higher CAS scores represented worse outcomes.

SECONDARY OUTCOMES:
muscle and retrobulbar fat volume change | 6 months after initiation of IVMP
  To compare the change in volume of extra-ocular muscles and retro bulbar fat after orbital radiotherapy, comparing standard with reduced-dose orbital radiotherapy
change in diplopia | 6 months after initiation of IVMP
  To compare the difference in prism deviation in primary gaze after standard and reduced-dose orbital radiotherapy
change in quality of life | 6 months after initiation of IVMP
  To compare the difference in Graves' ophthalmopathy quality of life (GO-QOL) scores (Thai version) between standard and reduced-dose orbital radiotherapy. The total QOL scores range from 0 to 100 with higher scores indicating a better health status.
Radiation toxicities | 6 months after initiation of IVMP
  To compare the summation of the Radiation Therapy Oncology Group (RTOG) toxicity scores (including dry eye, eye pain, keratitis, eyelid, conjunctiva, lacrimal gland, cornea, iris and skin toxicities) after standard and reduced-dose orbital radiotherapy. The RTOG gradings range from grade 0 to grade 4 in each item. The total toxicity scores range from 0-34, with a higher score indicating more severe side effects.
Visual acuity (VA) | 6 months after initiation of IVMP
  -To compare the differences in visual acuity (logMAR) change after standard and reduced-dose orbital radiotherapy
Visual field (VF) | 6 months after initiation of IVMP
  - To compare the differences of Humphrey's visual field (mean deviation) change after standard and reduced-dose orbital radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Janjira Petsuksiri, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkok Noi, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) may include sensitive information about participants, such as medical history or demographic details, particularly regarding their quality of life. Sharing IPD will be conducted in accordance with Siriraj Institutional Review Board (IRB) regulations for personal data protection."
Supporting Information: Study Protocol
Time Frame: April 15 2024- April 15 2028
Access Criteria: * Require researchers to demonstrate that their request for access to IPD has received ethical approval from Siriraj institution's Institutional Review Board (IRB).
  * Require researchers to provide a clear and specific purpose for requesting access to IPD, such as conducting further analysis, validation studies, or meta-analyses related to the research findings.
  * Require researchers to sign a data use agreement outlining the terms and conditions for accessing and using the IPD, including confidentiality, data security, and compliance with relevant regulations.
  * Request information about the researchers' plans for disseminating the findings obtained from the IPD, including intentions to publish or present the results in scientific journals, conferences, or other venues.
  * Consider requests from researchers interested in collaborating on future research projects or initiatives related to the research topic or dataset.

REFERENCES:
- [Result] Hoang TD, Stocker DJ, Chou EL, Burch HB. 2022 Update on Clinical Management of Graves Disease and Thyroid Eye Disease. Endocrinol Metab Clin North Am. 2022 Jun;51(2):287-304. doi: 10.1016/j.ecl.2021.12.004. Epub 2022 May 11. PMID 35662442
- [Result] San Miguel I, Arenas M, Carmona R, Rutllan J, Medina-Rivero F, Lara P. Review of the treatment of Graves' ophthalmopathy: The role of the new radiation techniques. Saudi J Ophthalmol. 2018 Apr-Jun;32(2):139-145. doi: 10.1016/j.sjopt.2017.09.003. Epub 2017 Sep 21. PMID 29942184
- [Result] Bartalena L, Kahaly GJ, Baldeschi L, Dayan CM, Eckstein A, Marcocci C, Marino M, Vaidya B, Wiersinga WM; EUGOGO dagger. The 2021 European Group on Graves' orbitopathy (EUGOGO) clinical practice guidelines for the medical management of Graves' orbitopathy. Eur J Endocrinol. 2021 Aug 27;185(4):G43-G67. doi: 10.1530/EJE-21-0479. PMID 34297684
- [Result] Marcocci C, Bartalena L, Bogazzi F, Bruno-Bossio G, Lepri A, Pinchera A. Orbital radiotherapy combined with high dose systemic glucocorticoids for Graves' ophthalmopathy is more effective than radiotherapy alone: results of a prospective randomized study. J Endocrinol Invest. 1991 Nov;14(10):853-60. doi: 10.1007/BF03347943. PMID 1802923
- [Result] Torres Royo L, Antelo Redondo G, Arquez Pianetta M, Arenas Prat M. Low-Dose radiation therapy for benign pathologies. Rep Pract Oncol Radiother. 2020 Mar-Apr;25(2):250-254. doi: 10.1016/j.rpor.2020.02.004. Epub 2020 Feb 22. PMID 32140081
- [Result] Abdus-Salam AA, Olabumuyi AA, Jimoh MA, Folorunso SA, Orekoya AA. The role of radiation treatment in the management of inflammatory musculoskeletal conditions: a revisit. Radiat Oncol J. 2020 Sep;38(3):151-161. doi: 10.3857/roj.2020.00178. Epub 2020 Jun 18. PMID 33012142
- [Result] Weissmann T, Lettmaier S, Donaubauer AJ, Bert C, Schmidt M, Kruse F, Ott O, Hecht M, Fietkau R, Frey B, Putz F. Low- vs. high-dose radiotherapy in Graves' ophthalmopathy: a retrospective comparison of long-term results. Strahlenther Onkol. 2021 Oct;197(10):885-894. doi: 10.1007/s00066-021-01770-9. Epub 2021 Apr 16. PMID 33860819
- [Result] Johnson KT, Wittig A, Loesch C, Esser J, Sauerwein W, Eckstein AK. A retrospective study on the efficacy of total absorbed orbital doses of 12, 16 and 20 Gy combined with systemic steroid treatment in patients with Graves' orbitopathy. Graefes Arch Clin Exp Ophthalmol. 2010 Jan;248(1):103-9. doi: 10.1007/s00417-009-1214-3. Epub 2009 Oct 29. PMID 19865824
- [Result] Kahaly GJ, Rosler HP, Pitz S, Hommel G. Low- versus high-dose radiotherapy for Graves' ophthalmopathy: a randomized, single blind trial. J Clin Endocrinol Metab. 2000 Jan;85(1):102-8. doi: 10.1210/jcem.85.1.6257. PMID 10634372
- [Result] Kim M, Chang JH, Lee NK. Quantitative analysis of extraocular muscle volume and exophthalmos reduction after radiation therapy to treat Graves' ophthalmopathy: A pilot study. Eur J Ophthalmol. 2021 Mar;31(2):340-345. doi: 10.1177/1120672119873841. Epub 2019 Sep 9. PMID 31496266
- [Result] Lumyongsatien M, Keeratidamkerngsakul B, Pornpanich K, Vangveeravong S, Saonanon P, Wiwatwongwana D, Mahaisavariya P, Aryasit O, Pongpirul K. Development and psychometric properties of the Thai Graves' ophthalmopathy quality of life (GO-QOL) questionnaire. J Patient Rep Outcomes. 2019 Dec 31;4(1):1. doi: 10.1186/s41687-019-0164-8. PMID 31893319

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT06392906/Prot_SAP_000.pdf